CLINICAL TRIAL: NCT05824923
Title: A Prospective, Multicenter, Randomized Controlled Trial to Evaluate the Safety and Efficacy of Single-use Ring-shaped Pulmonary Artery Radiofrequency (RF) Ablation Catheter and Pulmonary Artery RF Ablation Generator for the Treatment of Pulmonary Hypertension Associated With Left Heart Failure
Brief Title: A Trial to Evaluate the Safety and Efficacy of Pulmonary Artery Denervation for the Treatment of Pulmonary Hypertension Associated With Left Heart Failure
Acronym: PADN-HF-PH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pulnovo Medical (Wuxi) Co., Ltd. (Industry)
Collaborators: The General Hospital of Northern Theater Command (Other); The First Affiliated Hospital with Nanjing Medical University (Other); First Hospital of Tsinghua University (Other); Cangzhou Central Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Guangdong Provincial People's Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Tongji Hospital (Other); Second Hospital of Jilin University (Other); China-Japan Union Hospital, Jilin University (Other); Shanxi Cardiovascular Hospital (Other); RenJi Hospital (Other); Shanghai 10th People's Hospital (Other); Beijing Anzhen Hospital (Other); West China Hospital (Other); Sichuan Academy of Medical Sciences (Other); The First Affiliated Hospital of Soochow University (Other); TEDA International Cardiovascular Hospital (Other); Tianjin Medical University General Hospital (Other); Renmin Hospital of Wuhan University (Other); Zhongnan Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); Zhejiang University (Other); Shengjing Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Gansu Provincial Hospital (Other); Yanan Hospital of Kunming City (Unknown); First Affiliated Hospital of Chongqing Medical University (Other); Huaihe Hospital of Henan University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Affiliated Hospital of Nanchang University (Other); Hunan Provincial People's Hospital (Other); Tianjin Medical University Second Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pulnovo-CO-2022-01
Record Dates: First submitted 2023-01-10; First posted 2023-04-24 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Hypertension; Heart Failure With Reduced Ejection Fraction; Hypertension; Vascular Diseases; Cardiovascular Diseases; Heart Failure; Heart Failure With Preserved Ejection Fraction; Heart Failure With Mid Range Ejection Fraction
Keywords: Pulmonary Artery Denervation; Pulmonary Hypertension Due to Left Heart Disease; Heart Failure; pulmonary hypertension; left heart failure
MeSH Terms: conditions — Hypertension, Pulmonary; Hypertension; Vascular Diseases; Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Intervention Model Description: At the 12-months visit, participants in the control group who still meet the inclusion and exclusion criteria can choose to receive PADN procedure.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Artery Denervation (PADN) (Experimental): Patients in the PADN group will receive pulmonary artery denervation procedure.
  Interventions: Procedure: Pulmonary arterial denervation; Drug: Guideline-directed medical therapy (GDMT) for heart failure
- Guideline-directed medical therapy (GDMT) for heart failure (Active Comparator): Patients in the control group will take their baseline anti-heart failure medications at the original doses according to 2023 ESC Guidelines for heart failure, without any changes except when medically required. The anti-heart failure drugs treatment is consistent in both arms.
  Interventions: Drug: Guideline-directed medical therapy (GDMT) for heart failure

INTERVENTIONS:
Procedure: Pulmonary arterial denervation — Contrast pulmonary artery (PA) angiography will be performed to localize the pulmonary artery bifurcation level and calculate the PA diameter. Once the anatomy deemed acceptable, the radiofrequency ablation catheter will be introduced into ostium of the left PA and the distal bifurcation area of the main PA.
  The catheter will be manoeuvred within the PA to allow energy delivery in a circumferential manner to ensure that the electrodes are tightly in contact with the endovascular surface. About three ablations at 45-55 ℃ for 120 seconds each will be performed in ostium of the left PA and the distal bifurcation area of the main PA.
  For non-atrial fibrillation patients, dual antiplatelet therapy for 1 month after PADN is recommended. Patients with atrial fibrillation should continue new oral anticoagulants and patients who underwent metal valve replacement should continued oral warfarin anticoagulation according to guidelines, which could determined by the physician.
  Other Names: PADN
  Arms: Pulmonary Artery Denervation (PADN)
Drug: Guideline-directed medical therapy (GDMT) for heart failure — GDMT medication recommendation including:
  * Angiotensin-converting enzyme inhibitor (ACEI) or angiotensin-receptor blocker (ARB) or angiotensin receptor-neprilysin inhibitor (ARNI)
  * Beta-receptor blocker (BB)
  * Mineralocorticoid receptor antagonist (MRA)
  * Sodium-glucose co-transporter 2 (SGLT2) inhibitor
  * Diuretics
  The medication regimen (type and dosage) will be the investigator's discretion in accordance with the 2023 ESC Guidelines for Heart Failure. The type and dosage of all GDMT medications (except for diuretics) should remain unchanged through follow-up duration (at 12-month visit), unless the participant's conditions need adjust of GDMT regimens. Dosage and single or combination of diuretics are all left at physician's discretion.
  Other Names: GDMT medication for heart failure

SUMMARY:
It's a phase III, prospective, multicenter, randomized controlled trial to evaluate the safety and efficacy of the pulmonary artery denervation (PADN) for heart failure (HF) patients diagnosed with pulmonary hypertension associate with left heart disease (PH-LHD) by right heart catheterization.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) patients who have received guideline-directed medical therapy (GDMT) based on the 2023 ESC Guidelines for HF and have reached clinical stable, and diagnosed with PH-LHD by right heart catheterization, will be randomized to the PADN group or control group in a 1:1 ratio to receive PADN combined with HF GDMT or HF GDMT, respectively. After the 12-month follow-up visit is completed, participants in the control group who still meet the inclusion and exclusion criteria can also choose to receive PADN.

Approximately 264 participants will be enrolled at up to 39 centers in China and followed for 3 years. The safety and efficacy of the PADN system, including RF ablation catheter and generator will be evaluated by comparing the therapeutic effect of the PADN group and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, ≤75 years old;
2. Diagnosed with chronic heart failure for at least 3 months, and have received the GDMT pharmacological treatment based on the 2023 ESC Guidelines for Heart Failure for at least 1 month;
3. Clinically stable defined by

   1. No intravenous diuretics, inotropes or vasodilators for at least 1 month, and
   2. Systolic blood pressure (SBP) ≥ 100 and < 160 mmHg and resting heart rate (HR) ≥50 and <100 bpm (<110 bpm for atrial fibrillation) on the day of the procedure
4. New York Heart Association (NYHA) class II-IVa;
5. 6MWD ≥ 100 m and < 450 m;
6. NT-proBNP > 125 pg/mL (BNP > 35 pg/mL);
7. Hemodynamic indicators (RHC) :

   1. Mean pulmonary arterial pressure (mPAP) > 20 mmHg
   2. Pulmonary capillary wedge pressure (PCWP) >15 mmHg
8. Understand and be willing to sign informed consent, and be willing to follow the follow-up plan required by the protocol.

Exclusion Criteria:

1. Any of the following:

   1. Hypertrophic cardiomyopathy with left ventricular outflow tract obstruction or systolic anterior motion; pericardial disease; infiltrative or inflammatory myocardial disease; valvular stenosis of any of the 4 valves, or severe regurgitation of aortic and pulmonary valves, or active endocarditis; or
   2. Symptomatic carotid stenosis, or transient ischemic attack (TIA) or stroke within 30 days prior to randomization; or
   3. Untreated congenital heart disease; or
   4. Have received any revascularization, including coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) within 6 months prior to randomization; or anticipated to undergo coronary revascularization (CABG or PCI) within 6 months; or
   5. Artificial pacemakers, including single-chamber, dual-chamber and three-chamber pacemakers, have been implanted or are anticipated to be implanted within 6 months; or
   6. Anticipated to undergo ablation of atrial fibrillation within 6 months; or
   7. Anticipated to undergo heart valve surgery (valve replacement, valvuloplasty) within 6 months; or
   8. Listing for heart/heart-lung transplantation or anticipated to implant a ventricular assist device (VAD)
2. Other types of pulmonary hypertension, including WHO Group1, Group3, Group4, Group5;
3. Received pulmonary arterial hypertension (PAH) targeted drugs within 1 month prior to randomization;
4. Anticipated to undergo any surgery within 6 months;
5. The cardiac index (CI) of RHC < 1.5L/min/m²;
6. Severe renal insufficiency (eGFR <30mL/min/1.73m² by MDRD formula);
7. Severe liver insufficiency (Child-Pugh classification C);
8. Platelet count < 50 × 10^9/L;
9. Life expectancy <1 year;
10. Systemic inflammation or other disease requiring long-term use of glucocorticoids or immunosuppressants;
11. Active infection requiring oral or intravenous antibiotics;
12. Body mass index (BMI) >40 kg/m²;
13. Pregnant or lactating women, or plan to pregnant in one year;
14. Participated in other clinical trials within 3 months prior to signing the informed consent;
15. Any other circumstances that investigators deem inappropriate to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Worsening, defined as the occurrence of any of the followings: | immediately after the randomization to the last enrolled subject having at least 6 months follow-up
  1. Requiring intravenous medication (inotropes, diuretics or vasodilators) due to worsening of heart failure
  2. Rehospitalization due to heart failure
  3. 6MWD decreased by > 10% or > 30m compared with baseline
  4. Referral for heart/heart-lung transplantation
  5. All-cause death

SECONDARY OUTCOMES:
Parameters measured by transthoracic echocardiography(TTE) | 6 months, 1 year, 3 years
  Changes in left ventricular Tei index from baseline.
Parameters measured by transthoracic echocardiography(TTE) | 6 months, 1 year, 3 years
  Changes in left ventricular ejection fraction (LVEF) from baseline.
Parameters measured by transthoracic echocardiography(TTE) | 6 months, 1 year, 3 years
  Changes in left ventricular end-diastolic diameter (LVDd) from baseline.
Parameters measured by transthoracic echocardiography(TTE) | 6 months, 1 year, 3 years
  Changes in left ventricular end-systolic diameter (LVSd) from baseline.
Parameters measured by transthoracic echocardiography(TTE) | 6 months, 1 year, 3 years
  Changes in E/E' ratio from baseline.
Parameters measured by transthoracic echocardiography(TTE) | 6 months, 1 year, 3 years
  Changes in septum E' from baseline.
Parameters measured by transthoracic echocardiography(TTE) | 6 months, 1 year, 3 years
  Changes in lateral wall E' from baseline.
Parameters measured by transthoracic echocardiography(TTE) | 6 months, 1 year, 3 years
  Changes in left ventricular global longitudinal strain (LVGLS) from baseline.
N-terminal pro-B-type natriuretic peptide (NT-proBNP) | 6 months
  Changes in N-terminal pro-B-type natriuretic peptide (NT-proBNP) from baseline
6 minute walk distance(6MWD) difference from baseline | 6 months, 1 year, 3 years
  The 6MWD test was conducted according to the American Thoracic Society guidelines.
Changes in the Kansas City Cardiomyopathy Questionnaire(KCCQ) overall summary score from baseline | 1 month, 6 months, 1 year, 2 years, 3 years
  The KCCQ is a self-administered, 23-item questionnaire to provide a better description of quality of life in patients with heart failure. The overall summary score range from 0 to 100, higher score means higher quality of life.
Intravenous medication due to worsening of heart failure | 1 month, 6 months, 1 year, 2 years, 3 years
  Number of patients requiring intravenous medication (inotropes, diuretics or vasodilators) due to worsening of heart failure
Rehospitalization due to heart failure | 1 month, 6 months, 1 year, 2 years, 3 years
  Number of patients with rehospitalization due to heart failure
Heart/heart-lung transplantation | 1 month, 6 months, 1 year, 2 years, 3 years
  Number of patients referred for heart/heart-lung transplantation
All-cause death | 1 month, 6 months, 1 year, 2 years, 3 years
  Number of death due to any cause

OTHER OUTCOMES:
Safety Outcome: AESI | within 30 days after the procedure
  Adverse events of special interest (AESI), defined as complications occurring within 30 days after the procedure, include:
  1. Thrombosis and embolism
  2. Perforation or dissection of the pulmonary artery requiring surgical treatment
  3. Pulmonary aneurysm
  4. Pulmonary artery stenosis
  5. Hemoptysis requiring surgical treatment
  6. Recurrent laryngeal nerve injury
  7. Complications at puncture site (including pain, infection, bleeding, hematoma, etc.)
  8. All-cause death
  9. Endotracheal intubation
  10. Mechanical circulation support
  11. Permanent implantation of a pacemaker or defibrillator
Safety Outcome: AE and SAE | throughout the clincialtrial
  Adverse events (AE) and serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Principal Investigator — The General Hospital of Northern Theater Command
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China